CLINICAL TRIAL: NCT01970891
Title: Electrical Stimulation for the Relief of Freezing of Gait (FOG)
Brief Title: Electrical Stimulation for the Relief of Freezing of Gait (FOG) in Parkinson's Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, Gearoid O Laighin, Professor, National University of Ireland, Galway, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMES_PD_S_FOG
Record Dates: First submitted 2013-10-19; First posted 2013-10-28 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Parkinson's Disease
Keywords: Freezing of Gait; Gait; Comfort; Pain tolerance; Pain; Sensory threshold; Motor threshold; Pain threshold
MeSH Terms: conditions — Parkinson Disease; Pain

STUDY DESIGN:
Intervention Model Description: Sensory electrical stimulation for the amelioration of FoG through the continuous delivery of stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Freezing of Gait amelioration (Experimental): Effect of neuromuscular stimulation device will be assessed on Freezing of Gait amelioration
  Interventions: Device: neuromuscular stimulation device

INTERVENTIONS:
Device: neuromuscular stimulation device — Effect of neuromuscular stimulation device at specific muscle sites will be examined for freezing of gait amelioration.

SUMMARY:
Potential for electrical stimulation to ameliorate Freezing of Gait (FOG)

DETAILED DESCRIPTION:
The purpose of this study is to investigate the potential for an electrical stimulation intervention to ameliorate Freezing of Gait (FOG) and related gait disturbances in Parkinson's patients.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic Parkinson's Disease (PD) (UK, PD Brain Bank Criteria)
* A Hoehn and Yahr stage of 2 - 4
* Exhibiting Freezing of Gait or another gait abnormality in the ON state.
* An ability to mobilise independently with or without a walker or walking cane for the purpose of research when in the 'ON' state

Exclusion Criteria:

* A serious cognitive impairment (MMSE<24)
* Pregnant or currently involved in another clinical trial.
* Pacemakers
* On opioid or neuropathic pain medication

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Time in FoG PTF | At time of intervention (seconds)
  We hypothesise that the delivery of continuous sensory electrical stimulation will reduce the percentage of time in FoG.
Number of FoG episodes occurring | At time of intervention (seconds)
  We hypothesise that the delivery of continuous sensory electrical stimulation will reduce the Number of FoG episodes Occurring (NFO).

CONTACTS AND LOCATIONS:
Overall Officials: Gearóid Ó Laighin, PhD, Principal Investigator — National University of Ireland, Galway
Locations (1):
- Participants' home in the Mid-West region of Ireland, Limerick, Ireland